CLINICAL TRIAL: NCT06480370
Title: Optimization of Transcranial Motor Evoked Potentials in Supratentorial Surgeries
Acronym: MEPO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-D0039
Record Dates: First submitted 2024-06-24; First posted 2024-06-28 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Arm (Experimental): Application of TES at different stimulation circuits, with different stimulation parameters and recording montages.
  Interventions: Device: ISIS IOM System

INTERVENTIONS:
Device: ISIS IOM System — Application of TES at different stimulation circuits, with different stimulation parameters and recording montages.

SUMMARY:
This project aims to optimize the methodology to elicite transcranial motor evoked potentials in intraoperative neurophysiological monitoring of brain surgery. It includes accelerometer measurements and microscope video image to determine movement of the surgical field, making possible minimization of movement during brain stimulation.

DETAILED DESCRIPTION:
Background: During supratentorial brain surgery there is a risk of iatrogenic injury resulting in post-operative motor deficits. Intraoperative neurophysiological monitoring (IONM) can help surgeons avoid this outcome, while also expanding evidence of its prognostic and preventive benefit (1, 2). However, there are still pending issues, such as standardization of optimal methodologies for data acquisition and interpretation as well as technical improvement.

There are two main IONM strategies: mapping to localize nervous structures, and monitoring to provide real-time assessment of functional integrity (3). With respect to monitoring, muscle motor evoked potentials (MEPs) enable motor system assessment. They can be elicited by pulse train transcranial electric stimulation (TES) through scalp electrodes placed at standard 10-20 system sites (C1, C2, C3, C4, Cz-1cm, Cz+6cm), or at neuronavigation-guided scalp sites. The stimulation circuit consists of the user-selected anode and cathode sites chosen from the scalp electrodes (4). The stimulation parameters are user-selected pulse duration, interstimulus interval (ISI), number of pulses, and single train stimulation vs. double-train or multi-train facilitation. MEP threshold is the stimulation intensity required to elicit a certain number of MEPs with a predefined amplitude. The recording montage consists of user-selected recording electrode orientation and target muscles. Practitioner preferences for these technical aspects vary widely (5), and can influence monitoring efficacy.

During surgery, significant MEP deterioration from an earlier baseline indicates a warning based on various criteria such as amplitude reduction or threshold elevation (2). Warnings trigger rescue manoeuvres to recover MEPs. With reversible MEP deterioration (recovery to values above the warning level), a post-operative motor deficit might be prevented. Continuous real-time monitoring facilitates this favourable result by providing early warnings, and is therefore important. With irreversible MEP deterioration there is an increased risk of a motor deficit (1), and discontinuous intermittent monitoring may fail to help prevent this adverse outcome.

A major concern regarding TES MEPs is that the stimuli often produce movement of the surgical field, which entails the risk of the patient being harmed by surgical manoeuvres if they are not paused during the measurements (4). This can delay the surgical procedure and/or preclude real-time monitoring. Thus, there is a need to establish optimal TES MEP methodology that minimizes objectively assessed movement.

Objective: The hypothesis of this project is that MEP stimulation and recording paradigms can be optimized to minimize movement of the surgical field during supratentorial brain surgery. Consequently, the overall aim is to identify the most effective stimulation and recording techniques to maximize TES MEP performance by minimizing movement. The specific objectives are to determine:

1. The best stimulation circuit to elicit MEPs with the lowest possible movement;
2. The best stimulation parameters to elicit MEPs with the lowest possible movement;
3. The best recording montages to obtain MEPs with the lowest possible stimulation threshold.

Methods: General methods: Adult patients undergoing routine brain surgery with IONM and giving informed consent will be eligible. Muscle MEP recordings will be performed from limbs ipsilateral to the operation side. Patients with preoperative ipsilateral motor impairment will be excluded. Movement and MEP threshold will be the primary endpoints. Movement will be assessed through one accelerometer on the forehead (with quantification through kinetic energy). For comparison (secondary endpoint), another accelerometer on the ipsilateral shoulder to the recording site will be used, as well as the subjective evaluation by the surgeon on an ordinal scale, through visualization of the surgical field. Additionally, we propose to quantify the magnitude of motion using post-processing of digital images from the surgical microscope.

Comparative analyses of movement and MEP thresholds will be performed by successively varying one of the variables and keeping the others at Inselspital standard. Videos of the surgical field will be recorded with the microscope for all the proposed experimental setups, to recover the images for the quantification of the movement.

The study will be divided into four different parts, each of them with different steps (outlined below). Consequently, each patient participates in a specific part and stepThis subdivision is necessary due to time constraints in the operating room, as it would not be feasible to perform all the different combinations on every patient.

Patients who have already been included in the study and require a redo surgery will also be eligible for inclusion in a different part or step of the study.

Threshold current will be defined as the minimum current to elicit MEP responses with an amplitude higher than 20 µV in at least 5 consecutive trials. The procedure will be to increase current until MEPs appear, then reduce current until they disappear, and then finely adjust current to the minimum for a consistent response.

Part 1: determination of the best stimulation circuit. Step 1 - comparison of 10-20 system stimulation circuits: Evaluation of 12 patients. Circuits of C1/C2, C3/C4, and C3 or C4/Cz-1cm for upper limb MEPs, and C1/C2, C3/C4, and Cz-1cm/Cz+6cm for lower limb MEPs. Acquisition of 12 MEPs per limb with each circuit.

Step 2 - comparison of the best Step 1 circuit to the neuronavigation-guided stimulation circuit: Evaluation of 16 patients. Acquisition of 22 upper limb MEPs with each circuit.

Part 2: determination of the best stimulation parameters. Step 1 - comparison of different pulse durations: Evaluation of 21 patients. Pulse duration of 100, 200, 350, 500, 650, 800, and 1000 µs. Acquisition of 21 upper limb MEPs with each pulse duration.

Step 2 - comparison of different ISIs: Evaluation of 30 patients (15 per limb). ISI of 1, 2, 3, 4, and 5 ms. Acquisition of 20 upper and lower limb MEPs with each ISI.

Step 3 - comparison of different numbers of pulses: Evaluation of 15 patients. Number of pulses of 3, 4, 5, 7, and 9. Acquisition of 20 upper limb MEPs with each number of pulses.

Step 4 - comparison of single train to double-train facilitation at different inter train intervals (ITIs): Evaluation of 21 patients. Single train, double train (2/7 and 4/4 pulses). ITI of 20, 85, and 150 ms. Acquisition of 21 upper limb MEPs with each paradigm.

Step 5 - comparison of single train to multi-train facilitation at different rates: Evaluation of 21 patients. Single train at rate of 0.5 Hz. Multi-train facilitation at rates of 1, 2, 3, 4, 5, and 6 Hz. Acquisition of 21 upper limb MEPs with each paradigm.

Part 3: determination of the best recording montages. Step 1 - comparison of recording electrode orientations: Evaluation of 12 patients. Recordings from extensor digitorum communis (EDC) and tibialis anterior (TA). Three recording orientations: 1) bipolar perpendicular to muscle fibres, 2) bipolar parallel to muscle fibres, and 3) referential to the distal muscle tendon. Determination of threshold* per orientation within each muscle.

Step 2 - determination of muscles of choice in distal upper limbs: Evaluation of 21 patients. Recordings from abductor pollicis brevis (APB), abductor digiti minimi (ADM), first dorsal interosseous, EDC, flexor carpi radialis (FCR), APB/ADM, and EDC/FCR. Determination of threshold* for all muscles.

Step 3 - determination of muscles of choice in distal lower limbs: Evaluation of 18 patients. Recordings from abductor hallucis (AH), extensor digitorum brevis (EDB), TA, soleus, AH/EDB, and TA/soleus. Determination of threshold* for all muscles.

Part 4: Evaluation of 16 patients. Comparison of best stimulation and recording methodology from the results of Parts 1 to 3 with the current standard in our department. Acquisition of 22 MEPs per limb by paradigm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed by the subject
* The patient has a supra-tentorial lesion requiring surgery
* The patient is undergoing neurosurgery with the use of MEP monitoring during surgery to protect functional tissue* (During routine preparation for the surgery, patients are checked for any relative contraindications as listed in the user manual of the ISIS IOM System (see p. 11, chapter 2.2.4 of the user manual). Every relative contraindication must be weighed against the risk and benefits of the measurement signals which are routinely needed for the surgical intervention. There are no absolute contraindications for the ISIS IOM System.)
* The patient is older than 18 years

Exclusion Criteria:

* No need for MEP monitoring
* Vulnerable subjects (pregnant, impaired consciousness)
* People who do not want to participate in the study
* Emergency procedures in which no consent was obtained before the operation
* Multiple surgeries on the same patient
* Preoperative non-affected arm or leg motor deficit (MRC <5), that is to say, no motor deficit of the arm or leg ipsilateral to the surgery
* Inhalational anesthesia
* Persisting neuromuscular blockade
* Impossibility to place the stimulating or recording electrodes in the appropriate site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
threshold of stimulation and patient movement | during surgery
  threshold of stimulation and patient movement quantified by an accelerometer placed on the forehead of the patient

SECONDARY OUTCOMES:
patient movement | during surgery
  patient movement quantified by an accelerometer on the shoulder
subjective evaluation of magnitude of motion | end of surgery
  subjective evaluation by the surgeon of magnitude of motion using post-processing of digital images from the surgical microscope
quantification of magnitude | end of surgery
  quantification of magnitude of motion using post-processing of digital images from the surgical microscope

CONTACTS AND LOCATIONS:
Overall Officials: Seidel Kathleen, MD, Principal Investigator — Department of Neurosurgery
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holdefer RN, Skinner SA. Commentary : The value of intraoperative neurophysiological monitoring: evidence, equipoise and outcomes. J Clin Monit Comput. 2017 Aug;31(4):657-664. doi: 10.1007/s10877-016-9910-0. Epub 2016 Aug 1. PMID 27481235
- [Background] Asimakidou E, Abut PA, Raabe A, Seidel K. Motor Evoked Potential Warning Criteria in Supratentorial Surgery: A Scoping Review. Cancers (Basel). 2021 Jun 4;13(11):2803. doi: 10.3390/cancers13112803. PMID 34199853
- [Background] Seidel K, Beck J, Stieglitz L, Schucht P, Raabe A. The warning-sign hierarchy between quantitative subcortical motor mapping and continuous motor evoked potential monitoring during resection of supratentorial brain tumors. J Neurosurg. 2013 Feb;118(2):287-96. doi: 10.3171/2012.10.JNS12895. Epub 2012 Nov 30. PMID 23198802
- [Background] Macdonald DB, Skinner S, Shils J, Yingling C; American Society of Neurophysiological Monitoring. Intraoperative motor evoked potential monitoring - a position statement by the American Society of Neurophysiological Monitoring. Clin Neurophysiol. 2013 Dec;124(12):2291-316. doi: 10.1016/j.clinph.2013.07.025. Epub 2013 Sep 18. PMID 24055297
- [Background] Dulfer SE, Gadella MC, Sahinovic MM, Lange F, Absalom AR, Groen RJM, Szelenyi A, Drost G. Stimulation parameters for motor evoked potentials during intraoperative spinal cord monitoring. A systematic review. Clin Neurophysiol. 2023 May;149:70-80. doi: 10.1016/j.clinph.2023.02.170. Epub 2023 Mar 4. PMID 36924672
- [Background] Fujii M, Maesawa S, Motomura K, Futamura M, Hayashi Y, Koba I, Wakabayashi T. Intraoperative subcortical mapping of a language-associated deep frontal tract connecting the superior frontal gyrus to Broca's area in the dominant hemisphere of patients with glioma. J Neurosurg. 2015 Jun;122(6):1390-6. doi: 10.3171/2014.10.JNS14945. Epub 2015 Mar 27. PMID 25816090
- [Background] Kapsalakis IZ, Kapsalaki EZ, Gotsis ED, Verganelakis D, Toulas P, Hadjigeorgiou G, Chung I, Fezoulidis I, Papadimitriou A, Robinson JS, Lee GP, Fountas KN. Preoperative evaluation with FMRI of patients with intracranial gliomas. Radiol Res Pract. 2012;2012:727810. doi: 10.1155/2012/727810. Epub 2012 Jul 12. PMID 22848821
- [Background] Moiyadi A, Velayutham P, Shetty P, Seidel K, Janu A, Madhugiri V, Singh VK, Patil A, John R. Combined Motor Evoked Potential Monitoring and Subcortical Dynamic Mapping in Motor Eloquent Tumors Allows Safer and Extended Resections. World Neurosurg. 2018 Dec;120:e259-e268. doi: 10.1016/j.wneu.2018.08.046. Epub 2018 Aug 21. PMID 30138733
- [Background] Raabe A, Beck J, Schucht P, Seidel K. Continuous dynamic mapping of the corticospinal tract during surgery of motor eloquent brain tumors: evaluation of a new method. J Neurosurg. 2014 May;120(5):1015-24. doi: 10.3171/2014.1.JNS13909. Epub 2014 Mar 14. PMID 24628613
- [Background] Schucht P, Seidel K, Beck J, Murek M, Jilch A, Wiest R, Fung C, Raabe A. Intraoperative monopolar mapping during 5-ALA-guided resections of glioblastomas adjacent to motor eloquent areas: evaluation of resection rates and neurological outcome. Neurosurg Focus. 2014 Dec;37(6):E16. doi: 10.3171/2014.10.FOCUS14524. PMID 25434385